CLINICAL TRIAL: NCT04365985
Title: Study of Immunomodulation Using Naltrexone and Ketamine for COVID-19
Acronym: SINK COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of the decrease in COVID cases, enrollment is extremely low. Given the current study design, it is not possible to gather data necessary to answer the question about whether study treatment reduces mortality
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Matthew Sims, MD, PhD, Director Infectious Disease Research, Beaumont Health; Professor of Internal Medicine and Foundational Medical Studies, OUWB School of Medicine, Corewell Health East
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-097
Record Dates: First submitted 2020-04-26; First posted 2020-04-28 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome (SARS); Coronavirus Infections
Keywords: naltrexone; ketamine; cytokine storm; Interleukin-2; therapeutic treatment
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome; Coronavirus Infections; Cytokine Release Syndrome | interventions — Naltrexone; vivitrol; Ketamine; Sugars

STUDY DESIGN:
Intervention Model Description: Prospective, single center, randomized, double blinded study of naltrexone with an open label extension using ketamine as a rescue drug for patients who progress in their disease
Who Masked: Participant, Care Provider, Investigator
Masking Description: No other parties blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo by mouth 1 time per day for patients with stage I or stage 2A COVID-19
  Interventions: Other: Placebo
- Naltrexone (Experimental): Naltrexone 4.5 mg by mouth 1 time per day for patients with stage I or stage 2A COVID-19.
  Interventions: Drug: Naltrexone
- Ketamine (Experimental): Ketamine IV infusion (0.15 mg/kg based on total body weight for maximum 20 mg every 6 hours) for patients with stage 2B or stage 3 COVID-19; may be increased to 0.3 mg/kg based on total body weight for a maximum of 30 mg every 6 hours if needed. Patients entering this arm from the placebo or naltrexone arms remain on those medications as well.
  Interventions: Drug: Naltrexone; Drug: Ketamine; Other: Placebo

INTERVENTIONS:
Drug: Naltrexone — Low dose naltrexone, 4.5 mg by mouth, given from date of admission through time participant is stable for discharge for inpatient participants with mild/moderate COVID-19 infection stages. Naltrexone will continue for 1 month post hospital discharge. Patients progressing to requirement for advanced oxygenation will be reassess when sedation and assigned to Ketamine arm. Naltrexone may be reduced to 1.5 mg/day if interfering with sedation and can be held when sedation and symptoms of withdrawal is an issue..
  Other Names: ReVia; Vivitrol
  Arms: Ketamine; Naltrexone
Drug: Ketamine — Low dose ketamine hydrochloride given intravenously at a dosage of 0.15 mg/kg body weight for maximum 20 mg every 6 hours, to inpatient participants with advanced oxygenation requirements from either time of admission or time of progression of mild/moderate disease until time participant is stable for discharge, as a rescue treatment. If patient is transferred from the naltrexone or placebo arm, they will continue to receive naltrexone/placebo. Dosage of ketamine may be increased to 0.3 mg/kg body weight, maximum 30 mg every 6 hours, if participant does not respond at the lower dosage. Ketamine can be reduced back to 0.15 mg/kg at the clinical decision of the investigator and when patient has hypertensive emergency, the dose can be held until hypertensive emergency is controlled.
  Other Names: Ketalar
  Arms: Ketamine
Other: Placebo — Oral placebo, given from date of admission through time participant is stable for discharge for inpatient participants in mild/moderate COVID-19 infection stages. Placebo will continue for 1 month post discharge. Participants progressing to requirement for advanced oxygenation will be reassigned to Ketamine arm.
  Other Names: sugar pill
  Arms: Ketamine; Placebo

SUMMARY:
Ideal new treatments for Novel Coronavirus-19 (COVID-19) would help halt the progression disease in patients with mild disease prior to the need for artificial respiration (ventilators), and also provide a rescue treatment for patients with severe disease, while also being affordable and available in quantities sufficient to treat large numbers of infected people. Low doses of Naltrexone, a drug approved for treating alcoholism and opiate addiction, as well as Ketamine, a drug approved as an anesthetic, may be able to interrupt the inflammation that causes the worst COVID-19 symptoms and prove an effective new treatment. This study will investigate their effectiveness in a randomized, blinded trial versus standard treatment plus placebo.

DETAILED DESCRIPTION:
There is an urgent need to develop new treatments for Novel Coronavirus-19 (COVID-19) infection using easily available and affordable medications. We need to develop a treatment protocol which prevents progression of the disease and a treatment protocol to rescue those with advanced disease. In addition to anti-viral therapeutics currently under investigation in other trials, the addition of immunomodulators to the treatment regimen appears have to potential to act as agents which can reduce the pathogenicity of this disease by reducing the dysregulation of autoimmunity which is destructive of normal tissue and when unchecked rapidly leads to mortality.

COVID-19 infection has three stages and 80% of infected people stay in stage 1 or stage 2A (viral response and early pulmonary effects), however 20% of patients progress to stage 2B (late pulmonary effects), and of those about 20% progress to stage 3 (hyper-inflammation). An ideal treatment for COVID-19 would have a two-pronged strategy: a treatment that would slow or interrupt the progression of the disease from mild/moderate (stage 1-2A) to severe (stage 2B-3), and a treatment to rescue patients who have become severe. Promising data using tocilizumab, an monoclonal antibody targeting the cytokine Interleukin-6 (IL-6), suggests that interrupting IL-6 is one of the potential pathways to accomplish this.

Low-dose naltrexone has been used off-label for treatment of pain and inflammation in multiple sclerosis, Crohn's disease, fibromyalgia and other pain conditions. Lower than standard doses of naltrexone inhibit cellular proliferation of T- and B- cells and block Toll-like receptor 4 (TLR4), providing pain relief and anti-inflammatory benefit. Naltrexone at doses below the normal therapeutic dose appears to reduce production of multiple cytokines including IL-6 in a steady pace and is available as an oral preparation. As such it is ideal to use to attempt to modify progression to stage 2B as it can easily be given to both hospitalized patients and patients in the community.

Ketamine at low doses, below the normal anesthetic dose, appears to rapidly reduce the production of pro-inflammatory cytokines, especially IL-6 and tumor necrosis factor alpha (TNFα), for hours after an event which would induce the inflammatory response. This drug is given intravenously (IV), either by drip or push, and is easily given in a hospital environment. This could not easily be used in the community but could act as a rescue drug with lower cost and easier availability than tocilizumab, a monoclonal antibody targeting IL-6. Ketamine has been extensively studied in a variety of settings and indications with a well-established side-effect and dosing profile. Ketamine is generally well tolerated and remains inexpensive and widely available on the U.S. market and available for immediate use.

The trial will measure the ability of low dose naltrexone to reduce the progression of participants with COVID-19. In this study, naltrexone or placebo will be given to participants in early stages of COVID-19 infection in a randomized, double blinded manner, whereas the use of ketamine will be unblinded and given as a rescue agent should a participant progress. Additionally, should a participant be ineligible for the randomized portion of the study due to already being in a more advanced stage of the disease, they will be given the opportunity to enter the trial to receive ketamine without being randomized to naltrexone vs placebo.

Participants will continue to receive any standard of care COVID-19 treatment during their participation in this study. Laboratory blood tests such as IL-6 concentration, blood counts, liver and renal function panels as well as close physician supervision will be used to monitor participant condition during hospitalization. Participants will be contacted 1 month post discharge to evaluate outcomes and potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Positive for COVID -19
* Admitted to Beaumont Hospital - Royal Oak, Michigan
* Age ≥18
* Receiving ≤ 6 liters/minute oxygen by nasal cannula for randomization to either placebo or naloxone arm OR receiving ≥ 6 liters/minute oxygen by nasal cannula or requiring advanced oxygenation for placement in ketamine arm

Exclusion Criteria:

* Known allergy to naltrexone
* Known allergy to ketamine
* Diagnosis of schizophrenia or psychosis
* Pregnancy based on available medical history, existing labs, or verbal report
* On chronic high dose opioids > 90mg morphine mg equivalence
* Use of naltrexone or Vivitrol within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sims, MD PhD, Principal Investigator — Beaumont Health
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: Ketamine IV infusion (0.15 mg/kg maximum 20 mg every 6 hours) for patients with stage 2B or 3 COVID-19; may be increased to 0.3 mg/kg to a maximum of 30 mg every 6 hours if needed. Patients entering this arm from the placebo or naltrexone arms remain on those medications as well.
  Naltrexone: Low dose naltrexone, 4.5 mg by mouth, given from date of admission through time participant is stable for discharge for inpatients with mild/moderate COVID-19. Naltrexone will continue for 1 month post discharge. Patients progressing to requirement for advanced oxygenation will be reassessed and assigned to Ketamine arm. Naltrexone may be reduced to 1.5 mg/day if interfering with sedation .
  Placebo: Oral placebo, given from date of admission through time participant is stable for discharge for inpatient participants in mild/moderate COVID-19 infection stages. Placebo will continue for 1 month post discharge. Participants progressing to requirement for advanced oxygenation will be reassigned to Ketamine arm.
Period: Overall Study
Arm/Group | Placebo | Naltrexone | Ketamine
Started | 9 | 9 | 52
Completed | 9 | 9 | 52
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone | Ketamine | Total
Number analyzed (Participants) | 9 | 9 | 52 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.45 (16.29) | 68.52 (10.00) | 68.11 (13.20) | 67.82 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 18 | 26
  Male | 5 | 5 | 34 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 8 | 44 | 60
  Unknown or Not Reported | 1 | 1 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 10 | 14
  White | 6 | 7 | 32 | 45
  More than one race | 0 | 0 | 8 | 8
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 52 | 70

OUTCOME MEASURES:

1. Primary Outcome: Progression of Oxygenation Needs
Description: Count of participants initially presenting with mild/moderate disease who progress to requiring advanced oxygenation (high flow nasal canula, non-rebreather, continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), or intubation)
Time Frame: up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 9 | 52
Participants | 1 | 0 | 21

2. Secondary Outcome: Renal Failure
Description: Count of participants who develop or experience worsened renal failure as defined by RIFLE criteria, a 5-point scale where the categories are labeled: Risk-Injury-Failure-Loss-End stage renal disease, with Risk being the least severe and End stage renal disease being the most severe. The criteria for determination of stage are factors of serum creatinine and urine output. Numbers of participants worsening one or more RIFLE stages will be reported.
Time Frame: up to 1 month
Population: Missing data for 4 patients in Ketamine group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 9 | 48
Participants | 1 | 0 | 12

3. Secondary Outcome: Liver Failure
Description: Count of participants who develop or experience worsened liver failure as defined by serum transaminases five times normal limits
Time Frame: up to 1 month
Population: Missing data for 4 patients in Ketamine group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 9 | 48
Participants | 0 | 0 | 4

4. Secondary Outcome: Cytokine Storm
Description: Count of participants who develop cytokine storm as measured by elevated markers of inflammation (elevated D-dimer, hypofibrinogenemia, hyperferritinemia), evidence of acute respiratory distress syndrome (ARDS) measured by imaging findings and mechanical ventilator requirements, and/or continuous fever (≥ 38.1 ° Celsius unremitting)
Time Frame: up to 1 month
Population: Missing data for 4 patients in Ketamine group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 9 | 48
Participants | 0 | 0 | 0

5. Secondary Outcome: COVID Mortality
Description: Count of participants who die from COVID-19
Time Frame: up to 1 month post hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 9 | 52
Participants | 0 | 0 | 16

6. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay in days
Time Frame: up to 1 month
Population: Admission data not collected for Placebo and Naltrexone patients. Missing discharge data for 5 patients in ketamine group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 0 | 0 | 47
days |  |  | 21.37 (15.89)

7. Secondary Outcome: Intensive Care Unit (ICU) Admission
Description: Count of patients admitted to the ICU at any time during index hospitalization
Time Frame: up to 1 month
Population: Data not available for 1 patient in Naltrexone group and 5 patients in Ketamine group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 8 | 47
Participants | 2 | 1 | 28

8. Secondary Outcome: Intensive Care Unit (ICU) Duration
Description: Length of ICU stay in days
Time Frame: up to 1 month
Population: Patient in naltrexone group admitted to ICU had length of stay=0
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 2 | 1 | 28
days | 2.56 (0.71) | 0 (0) | 16.68 (11.25)

9. Secondary Outcome: Intubation
Description: Count of participants requiring intubation
Time Frame: up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 9 | 52
Participants | 0 | 1 | 29

10. Secondary Outcome: Intubation Duration
Description: Length of intubation, measured in days
Time Frame: up to 1 month
Population: No patients in Placebo group were intubated. For those intubated, data not available for 4 patients of 29 intubated in the Ketamine group
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 0 | 1 | 25
days |  | 3.32 (0) | 15.53 (14.12)

11. Secondary Outcome: Time Until Recovery
Description: Time measured in days from hospital admission to determination patient is stable for discharge
Time Frame: up to 1 month
Population: Patients not included who died during admission. Of 28 patients in ketamine group surviving to discharge, data missing for 5 patients. Of 8 patients in naltrexone group surviving to discharge, data missing for 1 patient.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Naltrexone | Ketamine
Number analyzed (Participants) | 9 | 7 | 23
days | 8.67 (5.79) | 8.71 (7.91) | 17.57 (22.14)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Systematic assessment of adverse events by review of medical records
Arm/Group | Placebo | Naltrexone | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/9 | 24/52
Serious Adverse Events (participants affected / at risk) | 4/9 | 9/9 | 52/52
Other Adverse Events (participants affected / at risk) | 9/9 | 7/9 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Naltrexone (N=9) | Ketamine (N=52)
ACUTE ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE CARDIAC ARREST DUE TO ARRYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE CARDIOPULMONARY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE CEREBRAL EDEMA AND ACUTE ENCEPHALOPATHY RELATED TO SUBACUTE INFARCT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ANEMIA REQUIRING TRANSFUSION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
ASPIRATION PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASYSTOLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
HEMORRHAGE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
CARDIOGENIC SHOCK SECONDARY TO ATRIAL FIBRILLATION WITH RAPID VENTRICULAR RESPONSE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIOPULMONARY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CRITICAL ILLNESS MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 6 (6)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA, EXTENDED-SPECTRUM BETA-LACTAMASE (ESBL) E COLI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL BLEED (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
HEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHAGIC SHOCK (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
HYPERKALEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
HYPOTENSION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
LABILE HYPOTENSION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
METHYCILLIN-RESISTANT STAPHLOCOCCUS AUREUS BACTEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OLIGOURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
PROGRESSION OF COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (10)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
SEPTIC SHOCK SECONDARY TO METHICILLIN-SUSCEPTIBLE STAPHYLOCOCCUS AUREUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEVERE METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SEVERE SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SHOCK (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
BACTEREMIA, STAPHLOCOCCUS EPIDERMIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
TOXIC METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
TRACHEAL EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
UNSTABLE ARRYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Naltrexone (N=9) | Ketamine (N=52)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
ALTERED MENTAL STATUS (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION WITH RAPID VENTRICULAR RATE (Cardiac disorders) | 1 (1) | 0 (0) | 5 (5)
BLEEDING (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 10 (10)
CHEST PAIN (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
CRITICAL ILLNESS MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4)
CYST, LOWER EXTREMITY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ELEVATED HEART RATE/BLOOD PRESSURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
EMESIS, ONE EPISODE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
EMESIS, FIVE EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
EPITAXIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
FEVER (General disorders) | 1 (1) | 0 (0) | 3 (3)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
LETHARGY, INCREASED (General disorders) | 1 (1) | 0 (0) | 0 (0)
MELENA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
PAIN, WRIST (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
XEROSTOMIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT04365985/Prot_SAP_000.pdf